CLINICAL TRIAL: NCT01914809
Title: Micro Array Analysis in Preeclampsia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2010-A00633-36; 2010-04 (Other: AP HM)
Record Dates: First submitted 2013-07-11; First posted 2013-08-02 (Estimated); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- group with a preeclampsia before 34 SA (Experimental)
  Interventions: Other: samples blood; Other: biopsy placentaire
- group with a normal pregnancy (Other)
  Interventions: Other: samples blood; Other: biopsy placentaire

INTERVENTIONS:
Other: samples blood
Other: biopsy placentaire

SUMMARY:
Preeclampsia is a frequent pathology. His etiology is doubtful.

Targets :

The study target is to identify a risk of preeclampsia group obtained with transcriptom analysis from circulating peripheric cells.

Design:

Multidisciplinary study (Gynaecology-Obstetric, Immunology, North CIC).

The study of the transcriptional history of peripheral blood cells of 2patients groups:

* A patient group with a preeclampsia before 34 SA
* A patient group with a normal pregnancy paired on main confusion factors. Blood sampling will be collected at the diagnosis and 8 weeks after delivery.

Results and perspectives

* Obtain a transcriptionnal signature of preeclampsia
* To identify new mechanism of the disease
* Identification of a specific transcriptom analysis with the comparison after delivery For long-term, the target is to identify risk patient in order to conduct easily preventive clinical trials in preeclamsia (primary prevention) and to consider a specific follow-up for risk patients.

ELIGIBILITY:
Inclusion Criteria:

* A prééclampsie (blood pressure superior to 140 mmHg and to 90 mmHg) and at least a cross of protein in the strip and/or more of 300mg / 24h after 20 LIMITED COMPANIES and before 34 limited companies.
* An informed consent signed by the patient will necessarily have to be obtained.
* Woman having been taken care during the pregnancy or at the time of the childbirth(delivery) by one of the participating teams to the current project.
* Caucasian Patient
* Wait primigeste and nullipare

Exclusion Criteria:

* Major Patient protected by the law.
* Patient deprived of freedom for administrative or judicial reasons.
* Patient not benefiting from a national insurance scheme.
* Refusal of the patient to participate in the study.
* Not Caucasian Patient
* Multipare Wait
* Multiple Pregnancy
* Existence of foetal deformation explaining a delay of growth or a foetal death in utero.
* Age 18 years and > 40 years.
* Absence of written consent or impossibility to receive the written consent (language or understanding).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-06-15 (Actual); Primary Completion 2021-01-25 (Estimated); Study Completion 2021-01-25 (Estimated)

PRIMARY OUTCOMES:
predictive markers of preeclampsia | 36 months
  blood samples

SECONDARY OUTCOMES:
analysis of placental transcriptional profile. | 36 months
  biopsie placentaire

CONTACTS AND LOCATIONS:
Overall Officials: LOIC MONDOLONI, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France